CLINICAL TRIAL: NCT04235257
Title: Immunogenicity of Fractional Dose of the Bivalent and Nonavalent Intradermal HPV Vaccines.
Brief Title: Intradermal, Fractional Dose of HPV Vaccines:
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Anna Wald, Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00008961
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: HPV Infection; HPV Vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bivalent HPV vaccine (Experimental): One-fifth fractional dose (0.1 ml) of bivalent HPV vaccine administered subcutaneously
  Interventions: Biological: HPV vaccine
- Nonavalent HPV vaccine (Experimental): One-fifth fractional dose (0.1 ml) of nonavalent HPV vaccine administered subcutaneously
  Interventions: Biological: HPV vaccine

INTERVENTIONS:
Biological: HPV vaccine — Gardasil 9 Bivalent HPV VLP Vaccine, one-fifth dose Nonavalent HPV VLP Vaccine, one-fifth dose

SUMMARY:
This randomized phase IV trial compares fractional dose of bivalent HPV vaccine to fractional dose of nonavalent HPV vaccine among men and women aged 27-45 years in Seattle, Washington. Participants will have immune response assessed at baseline, 4 weeks, 6 months, 12 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 27-45 years at enrollment
* Not intending to receive the HPV vaccine series for the duration of the study participation
* Willing and able to provide written informed consent, undergo clinical evaluation, and adhere to follow-up schedule

Exclusion Criteria:

* Prior immunization with HPV-vaccine (Cervarix, Gardasil-4, Gardasil-9)
* Currently pregnant or breastfeeding
* Immune deficiency or other immune disorder
* HIV infection or continued high risk for HIV; patients at risk for HIV who do not have a negative HIV test in the last 6 months will be excluded
* Cancer or chemotherapy (current, within 6 months, or anticipated in the future) except for fully excised non-melanoma skin cancer)
* Unstable medical condition (e.g., malignant hypertension, poorly controlled diabetes,
* Known allergy to vaccine components
* Prior history of HPV-associated cancer

Ages: 27 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV antibody detection after fractional HPV vaccination | 12 months
  HPV antibody response after delivery of a single, intradermal, fractional dose of the HPV-2 or HPV-9 vaccines

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No